CLINICAL TRIAL: NCT01135069
Title: Bioequivalence Study of Generic Tretinoin 0.1% Microsphere Gel, 0.1% Retin-A Micro® and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spear Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAM-01
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Generic (Active Comparator): treatment of acne for 12 weeks
  Interventions: Drug: Tretinoin microsphere 0.1%
- Brand (Active Comparator): Treatment of acne for 12 weeks
  Interventions: Drug: Brand Retin-A Micro tretinoin microsphere gel 0.1%
- Placebo (Placebo Comparator): Treatment if acne for 12 weeks as placebo
  Interventions: Drug: placebo microsphere gel

INTERVENTIONS:
Drug: Tretinoin microsphere 0.1% — Treatment of acne vulgaris
  Arms: Generic
Drug: Brand Retin-A Micro tretinoin microsphere gel 0.1% — Treatment of acne vulgaris
  Other Names: Retin-A Micro
  Arms: Brand
Drug: placebo microsphere gel — treatment of acne vulgaris
  Arms: Placebo

SUMMARY:
The objective will be to assess clinical bioequivalence of 0.1% Retin-A Micro® Gel and Spear Pharmaceutical's generic 0.1% Tretinoin Microsphere Gel with a placebo arm.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy male and female children and adult
* Written and verbal informed consent must be obtained. Patients age 12 to 17 (inclusive) must sign an assent for the study and a parent or a legal guardian must sign the informed consent.
* Women of child-bearing potential must be non-pregnant and non-nursing, and must be willing to avoid pregnancy during the course of the study and during the menstrual cycle following completion of their participation in the study.
* Able to refrain from the use of all other topical acne medications or antibiotics during the treatment period.
* Considered reliable and capable of understanding their responsibility and role in the study.

Exclusion Criteria:

* Significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hepatic, neurological, pancreatic, or renal disease.
* Abnormal pre-existing skin condition which might affect the normal course of acne vulgaris (e.g., eczema, psoriasis, albinism, or chronic vesiculobullous disorders).
* Use topical acne therapy during the two week period prior to study initiation.
* Use of systemic retinoid treatment within six months prior to study initiation.
* Pregnant or breast-feeding.
* Serious psychological illness.
* Participation in any clinical research study during the 30 day period preceding study initiation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krunal Patel, MD, Principal Investigator — Moore Clinical Research
Locations (1):
- Moore Clinical Research, Land O' Lakes, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Generic: Tretinoin Microsphere Gel 0.1%
- Brand: Retin-A Micro 0.1%
- Placebo: Microsphere Gel no active
Period: Overall Study
Arm/Group | Generic | Brand | Placebo
Started | 205 | 209 | 66
Completed | 169 | 177 | 56
Not Completed | 36 | 32 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic | Brand | Placebo | Total
Number analyzed (Participants) | 205 | 209 | 66 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 100 | 33 | 233
  Between 18 and 65 years | 105 | 109 | 33 | 247
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (7.4) | 21 (8.1) | 19 (6.7) | 21 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 150 | 42 | 342
  Male | 55 | 59 | 24 | 138
Region of Enrollment [Number; unit: participants]
  United States | 205 | 209 | 66 | 480

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Acne
Description: Counting of acne lesions both inflammatory and non-inflammatory
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Generic: treatment of acne for 12 weeks
  Percent change (reduction) in acne lesions was 74% reduction.
- Brand: Treatment of acne for 12 weeks
  Percent change (reduction) in acne lesions was 76% reduction
- Placebo: Treatment of acne for 12 weeks
  Percent change (reduction) in acne lesions was 58% reduction
Arm/Group | Generic | Brand | Placebo
Number analyzed (Participants) | 205 | 209 | 66
Percent change | -74 (.05) | -76 (.04) | -58 (.03)

ADVERSE EVENTS:
Arm/Group | Generic | Brand | Placebo
Serious Adverse Events (participants affected / at risk) | 0/205 | 0/209 | 0/66
Other Adverse Events (participants affected / at risk) | 26/205 | 29/209 | 10/66
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic (N=205) | Brand (N=209) | Placebo (N=66)
Irritation (Skin and subcutaneous tissue disorders) | 26 (26) | 29 (29) | 10 (10) — Tretinoin produces irritation

LIMITATIONS AND CAVEATS:
No unexpected problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other